CLINICAL TRIAL: NCT02449798
Title: A Prospective Feasibility Trial of AccuCath 2.25" BC Intravascular Catheter System With Retractable Coiled Tip Guidewire Placed in Difficult Access Patients in the Emergency Department
Brief Title: Prospective Feasibility Trial of AccuCath 2.25" Blood Control (BC) Placed in Difficult Access Patients in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VPW-STP-00007
Record Dates: First submitted 2015-05-16; First posted 2015-05-20 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Vascular Access Complication
Keywords: Difficult IV access; AccuCath; IV outcomes; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AccuCath 2.25" BC Intravascular Catheter (Experimental): Use of AccuCath 2.25" BC peripheral IV device for difficult IV access in emergency room patients who have had 2 previous attempts, identified as difficult IV access from patient history or non-palpable, non-visible veins.
  Interventions: Device: AccuCath 2.25" BC Intravascular Catheter

INTERVENTIONS:
Device: AccuCath 2.25" BC Intravascular Catheter — Long peripheral IV catheter designed for difficult IV access patients requiring deeper vessel access, often used with ultrasound guidance.
  Other Names: AccuCath; AccuCath peripheral IV; AccuCath IV device; AccuCath catheter system

SUMMARY:
Study objective is to evaluate user preference, time for procedure, insertion success rates, complications, completion of therapy and dwell time of the AccuCath 2.25" BC device placed in difficult IV access patients in the emergency department.

DETAILED DESCRIPTION:
A one arm, prospective feasibility study using the AccuCath 2.25" BC Intravascular Catheter System placed in the upper arm with ultrasound guidance, and the lower arm with and without ultrasound guidance based on clinical assessment. Subjects will be subjected to a maximum of 4 attempts. If unsuccessful by the 4th attempt, alternatives will be considered as per current standard of care.

Currently multiple IV attempts are made in difficult IV access patients without success. Patients are often escalated to more invasive lines due to the need for longer catheters without clinical indication. The study will evaluate the feasibility of AccuCath 2.25" BC as a low risk, lower cost alternative for this patient population in lieu of using a midline, peripherally inserted central line or central venous catheter when not clinically required for purposes of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > 18 years old;
2. Capable and willing to give informed consent;
3. English speaking;
4. Acceptable candidate for an elective, non-emergent peripheral IV as determined by ordering physician;
5. Admitted to inpatient area for minimum of 24 hours, preferably for average hospital length of stay;
6. Difficult venous access patient as defined by either 2 failed initial attempts without ultrasound guidance or a history of difficult access plus the inability to directly visualize or palpate a target vein.

Exclusion Criteria:

1. Male or female, < 18 years old;
2. Requirement for emergent IV placement (patient's condition would be compromised if there is a delay in IV placement);
3. Previous venous grafts or surgery at the target vessel access site;
4. Subjects with lymphedema or status-post mastectomy on affected side;
5. Currently involved in other investigational clinical trials (unless permission is granted by other study PI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Raio, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore - Long Island Jewish Health System, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AccuCath 2.25" BC Intravascular Catheter: Use of AccuCath 2.25" Blood Control (BC) peripheral intravenous (PIV) device for difficult IV access in emergency room patients who have had 2 previous attempts, identified as difficult IV access from patient history or non-palpable, non-visible veins.
  AccuCath 2.25" BC Intravascular Catheter: Long peripheral IV catheter designed for difficult IV access patients requiring deeper vessel access, often used with ultrasound guidance.
Period: Overall Study
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: Year] | 56.5 (19.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 41
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 55
  Black | 47
  Latino | 11
  Asian | 6
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: First Attempt Success Rate
Time Frame: At initial IV insertion attempt, generally from 3-15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Number analyzed (Participants) | 120
Participants | 92

2. Primary Outcome: Number of Catheter Attempts Required to Complete Successful PIV Placement
Time Frame: At IV insertion attempt, generally from 3-15 minutes
Measure: Median (Full Range); unit: Number of Catheters
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Number analyzed (Participants) | 120
Number of Catheters | 1 [1 to 3]

3. Secondary Outcome: Time to Catheter Placement
Description: Time will be measured from initial vessel insertion through successful cannulation
Time Frame: At initial IV insertion attempt through successful cannulation, generally from 3-15 minutes
Measure: Median (Full Range); unit: minutes
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Number analyzed (Participants) | 114
minutes | 2 [0 to 30]

4. Secondary Outcome: Complications
Description: Count of IV complications that require IV removal before completion of therapy. Includes infiltration, extravasation, phlebitis, occlusion, dislodgement, infection, leaking at site, pain at site
Time Frame: During IV dwell from initial insertion success through IV removal, usually ranges from 7-14 days but could be up to 29 days
Population: The total number of complications resulting from all 120 IV placement procedures is reported.
Measure: Number; unit: Complications
Units Other Than Participants: IV procedures
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Number analyzed (Participants) | 120
Number analyzed (IV procedures) | 120
Complications | 18

5. Secondary Outcome: Dwell Time
Description: IV dwell time in hours until IV is no longer needed or complicates.
Time Frame: Duration of IV dwell from initial insertion success through IV removal, usually ranges from 0-336 hours (0-14 days) but could be up to 696 hours (29 days)
Population: Admitted patients
Measure: Median (Full Range); unit: hours
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Number analyzed (Participants) | 85
hours | 90.98 [1.6 to 535.8]

6. Secondary Outcome: Completion of Therapy
Description: Count of whether the catheter lasted for the duration of intended therapy without complication requiring early removal.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Number analyzed (Participants) | 120
Participants | 102

7. Secondary Outcome: Patient Satisfaction
Description: A 5-point Likert scale (1-5) was used for measurement of satisfaction with overall IV insertion experience. A score of 1 indicated the lowest satisfaction, while a score of 5 indicated the highest satisfaction. A score of 3-5 was considered positive.
Time Frame: At end of IV insertion, first 3-15 minutes of procedure
Measure: Median (Full Range); unit: units on a scale
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Number analyzed (Participants) | 120
units on a scale | 5 [1 to 5]

8. Secondary Outcome: Patient Satisfaction
Description: A 5-point Likert scale (1-5) was used for measurement of satisfaction with overall IV performance at IV removal. A score of 1 indicated the lowest satisfaction, while a score of 5 indicated the highest satisfaction. A score of 3-5 was considered positive.
Time Frame: at IV removal, which can be up to a maximum of 29 days
Measure: Median (Full Range); unit: units on a scale
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Number analyzed (Participants) | 120
units on a scale | 5 [1 to 5]

9. Other Pre Specified Outcome: Number of Attempts Prior to AccuCath 2.25" Use
Description: Count of catheter attempts during initial insertion before patient identified as difficult IV access
Time Frame: Number of IV attempts made before patient identified as difficult access and enrolled in study, could range from 3-30 minutes during initial procedure attempts
Measure: Median (Full Range); unit: number of attempts
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Number analyzed (Participants) | 120
number of attempts | 3 [0 to 12]

ADVERSE EVENTS:
Time Frame: Treatment emergent anticipated and unanticipated serious and non-serious adverse events were recorded from catheter insertion until catheter removal. Catheter dwell time usually ranges from 0-336 hours (0-14 days) but could be up to 696 hours (29 days).
Description: The number and proportion of subjects in the Safety Patient Set reporting any given adverse event were tabulated according to the worst severity reported during the study period.
Arm/Group | AccuCath 2.25" BC Intravascular Catheter
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 6/120
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AccuCath 2.25" BC Intravascular Catheter (N=120)
Infiltration (Product Issues) | 6 — Infiltration results when the IV catheter is dislodged and fluid infuses into the tissue. It is characterized by edema, pallor, decreased skin temperature around the site, and pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No